CLINICAL TRIAL: NCT03686826
Title: Feasibility and Reliability of Multimodal Evoked Potentials
Acronym: EP-B
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01099; me16Fuhr2
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: evoked potentials (EP); motor evoked potentials (MEP); Somato-sensory evoked potentials (SSEP); multimodal evoked potentials (mmEP)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis patients
  Interventions: Procedure: Acquisition of MEP und SSEP
- healthy volunteers
  Interventions: Procedure: Acquisition of MEP und SSEP

INTERVENTIONS:
Procedure: Acquisition of MEP und SSEP — Acquisition of MEP und SSEP at two different time points within 1 to 30 days

SUMMARY:
Multimodal Evoked potentials (mmEP) reflect disease course of multiple sclerosis (MS) and are potentially suited as a biomarker for disease progression.

The acquisition of evoked potentials (EP) in this observatory trial is to evaluate the feasibility and test-retest reliability of motor and somato-sensory EP (MEP and SSEP) in an international multicenter setting in healthy subjects and subjects with multiple sclerosis (MS).

DETAILED DESCRIPTION:
Multimodal EP (mmEP) is being developed as a predictive biomarker to determine the clinical response to therapy. MEP and SSEP contributes significantly to the predictive value of mmEP. The variability of MEP and SSEP has limited its use in multicenter clinical trials. Recent technological advances and standardization of procedures has decreased the variability. The objective of this study is to evaluate the reliability of MEP and SSEP and feasibility of performing MEP and SSEP in an international, multicenter setting. Establishment of the reliability and feasibility of MEP and SSEP will allow for further development of this predictive biomarker in future clinical trials.

ELIGIBILITY:
Inclusion Criteria (Healthy controls):

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Have no significant health issues, ie neuropathy or other demyelinating disorder that can affect testing.

Inclusion Criteria (Patients with MS):

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations
* Diagnosis of MS (all types) with an expanded disability status scale (EDSS) 0.0 to 6.5
* Have measurable responses on both MEP and SSEP in at least one upper and one lower limb on visit 2. The MEP and SSEP responses do not need to be in the same limb
* Have no comorbid condition (ie neuropathy) that could affect testing

Exclusion Criteria:

* Inability to comply with study requirements
* Unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment
* Any diseases (e.g., non-MS demyelinating diseases), with the exception of diagnosis MS for the MS Cohort, that in the opinion of the Investigator, could influence evoked potential results (including but not limited to medullary trauma, morbid obesity, limb amputation, diabetes, other polyneuropathy)
* Conditions interfering with magnetic stimulation (including but not limited to epilepsy, movable metal implants in the body such as pacemakers or stents)
* MS relapse within 3 months of either sessions
* Initiation of treatment or dose adjustment within 1 month of either sessions with 4-Aminopyridin, Carbamazepine, Baclofen, Tizianid
* Febrile illness within 3 days of either sessions.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with MS will be recruited from the outpatient clinic at the University Hospital Basel as consecutive ongoing recruitment through project leader and Co-workers in daily clinical practice.
  Healthy subjects will be recruited by bulletin on notice-boards in the hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
intraclass correlation coefficient (ICC) of MEP and SSEP | time between Visit 1 (= Baseline = Day 0) and Visit 2 (= 1 day to 30 days after Visit 1)
  The primary analysis will be a descriptive statistical summary of MEP and SSEP results at the first session, the second session and overall. Intraclass correlation coefficients (ICC) will be calculated to assess the test-retest reliability between consecutive measurements and the interrater reliability between raters.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof. Dr. MD, Principal Investigator — University Hospital Basel; Department of Neurology
Locations (1):
- Dep. of Neurology, Hospital of the University of Basel, Basel, Switzerland